CLINICAL TRIAL: NCT05360706
Title: A Phase I/IIb Extension Study Assessing the Long-term Safety and Efficacy of an Adeno-associated Viral Vector Containing a Codon-optimized Human Factor IX Gene (AAV5-hFIX) Previously Administered to Adult Patients With Severe or Moderately Severe Haemophilia B During the CT-AMT-060-01 Phase I/II Study
Brief Title: Study of AAV5-hFIX in Severe or Moderately Severe Haemophilia B
Status: Active, not recruiting | Type: Observational
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: CSL220_1002 (CT-AMT-060-04); 2020-000739-28 (EudraCT Number)
Record Dates: First submitted 2022-04-26; First posted 2022-05-04 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — After biological samples have been analyzed, they will remain stored for potential re-analysis at any time during the study to a maximum of up to 1 year after the study has been completed, before being destroyed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CSL220: AAV5 containing a codon-optimized human factor IX gene
  Interventions: Genetic: AAV5-hFIX

INTERVENTIONS:
Genetic: AAV5-hFIX — AAV5 containing a codon-optimized human factor IX gene
  Other Names: CSL220

SUMMARY:
This is an open-label, extension study enrolling patients who have successfully completed all assessments in Study CT-AMT-060-01 (Years 1-5). Assessment phase will begin at Visit 36 (the first clinical visit in this extension study, approximately 5.5 years after the initial dosing visit Study CT-AMT-060-01) and go to Visit 45 (10-years post-dosing in Study CT-AMT-060-01).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with congenital hemophilia B who completed Study CTAMT-060-01
* Able to provide informed consent following receipt of verbal and written information about the trial.

Exclusion Criteria:

* Enrolled subjects will have already been assessed based on the exclusion criteria for Study CT-AMT-060-01.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male subjects with severe or moderately severe haemophilia B, who previously received an infusion of AMT-060 and completed all assessments in Study CTAMT-060-01
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse events Possibly or probably related to previous AAV5-hFIX administration | 6-10 years after dosing in CT-AMT-060-01 study
Neutralizing FIX antibodies (FIX inhibitors) | 6-10 years after dosing in CT-AMT-060-01 study
ALT/AST levels | 6-10 years after dosing in CT-AMT-060-01 study
Liver pathology score Assessed by ultrasound every 6 months | 6-10 years after dosing in CT-AMT-060-01 study
Alfa fetoprotein levels | 6-10 years after dosing in CT-AMT-060-01 study

SECONDARY OUTCOMES:
Endogenous Percent FIX activity | 6-10 years after dosing in CT-AMT-060-01 study
Total Consumption of FIX Replacement Therapy on-demand and prophylactic | 6-10 years after dosing in CT-AMT-060-01 study
Annualized bleeding rate Including all bleeds (treated and untreated), spontaneous bleeds, traumatic bleeds and joint bleeds | 6-10 years after dosing in CT-AMT-060-01 study
Number of Procedures (including major and minor surgeries) | 6-10 years after dosing in CT-AMT-060-01 study
Quality of Life questionnaire SF-36 score | 6-10 years after dosing in CT-AMT-060-01 study
Quality of Life questionnaire EQ-5D-5L score | 6-10 years after dosing in CT-AMT-060-01 study
Hemophilia Joint Health Score | 6-10 years after dosing in CT-AMT-060-01 study

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (6):
- Germany (2):
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Universitaetsklinikum Frankfurt - Klinikum der Johann Wolfgang Goethe Universitaet, Frankfurt
- Netherlands (4):
  - Amsterdam UMC - Locatie AMC, Amsterdam
  - Groningen UMC, Groningen
  - Erasmus MC, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.